CLINICAL TRIAL: NCT06285838
Title: Impact of Measures Taken to Contain COVID-19 on Hospital Surgical Care Services and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Singapore Health Services (Other)
Responsible Party: Principal Investigator, Sean Shao Wei Lam, Deputy Director, Singapore Health Services
Other Study IDs: 2020/2706
Record Dates: First submitted 2024-02-28; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: impact of measures; hospital surgical care services
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Swift and decisive actions on the part of healthcare and hospital authorities are required to effectively contain the current COVID-19 pandemic. These measures firstly allow personnel and facilities leeway to provide surge capabilities to meet anticipated increased demands on the healthcare service. In addition, by deferring none urgent hospital visits, admissions and investigations, such measures support social distancing and aid attempts to control disease transmission. Deferring perceived non-urgent patient services may however lead to unintended delayed diagnoses and exacerbation of current patient conditions and lead to increased emergency admissions and surgeries.

A policy decision was made that essential surgical services pertaining to cancer and urgent cardiovascular surgery were allowed but that surgeons had the option to postpone what is assessed to be less urgent cases. Increasingly patients also postpone their surgeries or visits because of anxieties over the developing situation. Elective surgical services at the Outram Campus were thus significantly reduced from January 2020 as part of the measures to contain the COVID-19 outbreak.

The surgical philosophy during this period was that a judicious policy that allowed surgeons to proceed with surgery deemed critical but to postpone those deemed less so will at the system level, avoid poor outcomes for patients who required surgery and yet successfully re-allocate resources required to address the unfolding pandemic.

DETAILED DESCRIPTION:
Cohort of patients who were treated will be analysed via retrospective medical records review. These patients are classified according to the institution, type of surgical procedures, the medical condition and the dates of surgical treatment. The study will be compared across four time periods as listed:

-1Jan-31Dec2020 -1Jan-31Dec2019 -1Jan-31Dec2018 -1Jan-31Dec2017

The study focus on surgical indices for selected high-volume cancer and non-cancer diagnoses over the period 1st January 2020 to 31 December 2020 and compare them with similar indices across the same period of time in the preceding 3 years in particular, for the following surgical procedures:

1. Surgeries for the following cancer diagnoses:

   1. breast cancer, [XIV- N60, no malignancy], [Malignant, II Neoplasms- C50], colorectal cancer, [C18, 19, 20],
   2. hepatocellular carcinoma, [C22]
2. Selected non-cancer surgeries: a. Cholecystectomy b. Abdominal hernia repair

ELIGIBILITY:
Inclusion Criteria:

* Patients who had the following surgeries during the period 01 Jan 2017 to 31 December 2020.

From the identified surgical procedure type as shown Surgeries for the following cancer-related procedures.

1. Breast Cancer
2. Colon Cancer
3. Liver
4. Rectum

Selected non-cancer surgeries.

1. Abdominal Wall
2. Gall bladder

Patients from SGH and its releated institute NCC Only local Singapore citizens

Exclusion Criteria:

No exclusion criteria

-

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients coming to SGH for surgeries
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Impact of measures taken to contain COVID-19 on hospital surgical care services and clinical outcomes | 4 years
  Study seeks to assess the effect of the measures taken to contain COVID 19 on patients who need surgical services measured by patient outcomes, such as, length of hospital stay (LOS), ICU stay, APACHE score, stage of cancer at surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Health Services Pte ltd, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazingi D, Navarro S, Bobel MC, Dube A, Mbanje C, Lavy C. Exploring the Impact of COVID-19 on Progress Towards Achieving Global Surgery Goals. World J Surg. 2020 Aug;44(8):2451-2457. doi: 10.1007/s00268-020-05627-7. PMID 32488665